CLINICAL TRIAL: NCT06012487
Title: Correlates and Control of Blood Pressure Variability
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Ebinger, Assistant Professor of Cardiology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY02827
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure Variability

STUDY DESIGN:
Intervention Model Description: This is a feasibility study of the feasibility of helping physicians select a protocol to reduce BPV in hypertensive patients on antihypertensive therapy. The duration of the study for Aim 2 is 2 visits, the first with a 48 hour ABPM and the second for a repeat 48 hour ABPM following any changes made at the discretion of the treating provider.
  The optional sub-study is also a feasibility study, designed to demonstrate the ability to simultaneously capture ABPM and SKNA data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambulatory Blood Pressure Monitor (ABPM) (Other): Participants on antihypertensive pharmacotherapy in the highest decile of BPV will be offered enrollment based on inclusion/exclusion criteria. Patient's will undergo a 48 hour ABPM to determine baseline BPV. Next, each patient's primary care physician will be guided through titrations to antihypertensive medications to a low BPV regimen (Amlodipine and Indapamide, with doses titrated to reach target blood pressure). Following this, patients will undergo repeat 48h ABPM to evaluate change in BPV. All medication decisions will be at the ultimate discretion of the treating physician.
  The optional sub-study will test the hypothesize that ABPM and SKNA data can be simultaneously captured and that BPV will be positively correlated with SKNA. Participants who enroll in the optional sub-study will be fitted with a single patch ECG which will capture high-fidelity ECG tracings from which SKNA can be determine in post-test analysis.
  Interventions: Drug: Low BPV Regimen

INTERVENTIONS:
Drug: Low BPV Regimen — Each the patients' physician will invite patients to complete a 48-hour ABPM, then undergo cross-titration from their current antihypertensive regimen to a low BPV regimen, consisting of Amlodipine and Indapamide. Study staff will suggest to the treating physician to initially start patients on Amlodipine 5mg daily, with uptitration to 10mg daily to a goal systolic blood pressure (SBP)<130 mmHg. Indapamide will be suggested to be added at 1.25mg daily and increased to 2.5mg daily, as needed to meet target SBP. Other antihypertensive medications will be suggested to be discontinued as the SBP target is reached. Patients not meeting target SBP on maximally tolerated Amlodipine and Indapamide will be suggested to have a long acting angiotensin-converting enzyme (ACE)/ angiotensin receptor blocker (ARB) added to their therapy. Patients will complete another 48-hour ABPM after 1 week at target SBP on the low-BPV regimen.

SUMMARY:
The purpose the research is to prospectively demonstrate agreement between EHR and ambulatory blood pressure monitor (ABPM) derived blood pressure variability (BPV), as well as the feasibility of reducing BPV using a data-driven pharmacotherapeutic approach. To this end, this is a feasibility study that will make use of the Cedars-Sinai Health System including the Medical Delivery Network and the clinics of all practitioners who use the same EHR.

DETAILED DESCRIPTION:
The primary research procedures are: assessment of blood pressure variability (BPV) using ABPM compared to EHR derived values; and to assess feasibility of a data driven pharmacotherapy intervention to reduce BPV among high BPV patients. As part of an option sub-study, participants may wear a single lead ECG patch to record skin sympathetic nerve activity (SKNA), which has been previously correlated with changes in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included.
* Patients followed continuously at Cedars-Sinai for at least 5 years, defined as at least 1 outpatient visit with a Cedars-Sinai physician at which a blood pressure was measured each of the last 2 calendar years
* Patients with a PCP in the Cedars-Sinai Medical Group or faculty practice
* Patients on antihypertensive therapy other than a DPH-CCB or thiazide-like diuretic
* Patients in the highest decile of BPV based on extracted BP data from the EHR

Exclusion Criteria:

* Any records flagged "break the glass" or "research opt out."
* Pregnant or breastfeeding patients (due to guideline recommendations for specific medications for the treatment of hypertension during pregnancy and breastfeeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure Variability | 48 hours
  Change in Average Real Variability from pre-intervention 48h Ambulatory Blood Pressure Monitor (ABPM) and post-intervention 48 ABPM

IPD SHARING:
Plan to Share IPD: No